CLINICAL TRIAL: NCT01012583
Title: Optical Coherence TomOgraphy Assessment of the Excel Drug-Eluting Stent With BiodegradablE polymeR vs. the Cypher Drug-Eluting Stent With Permanent Polymer
Brief Title: Optical Coherence TomOgraphy Assessment of the Drug-Eluting Stent
Acronym: OCTOBER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Chinese PLA General Hospital,Beijing,China, Chinese PLA General Hospital,Beijing,China
Other Study IDs: OCT-001
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Atherosclerosis
Keywords: Optical coherence tomography; Drug eluting stent; Biodegradable polymer; Intimal; Coverage; assess intimal hyperplasia of drug eluting stent with biodegradable polymer
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
BACKGROUND Treatment of coronary atherosclerotic disease has been significantly advanced by interventional cardiology, and the advent of coronary arterial stents. In comparison to angioplasty alone, stents have reduced the incidence of angiographic as well as clinical restenosis, the recurrence of angina, the need for coronary arterial bypass graft (CABG) surgery, repeat revascularization and the occurrence of major adverse cardiac events (MACE).However the long-term success of this therapy has been limited by the occurrence of in-stent restenosis. Despite the effectiveness of intracoronary stents in maintaining a larger luminal diameter, as compared to angioplasty alone, in-stent restenosis occurs within 6 to 9 months after stent placement in 15% to 35% of patients. While stents can reduce restenosis by blocking vascular recoil and remodeling, mechanical intervention alone has been incapable of treating this biological problem of neointimal hyperplasia, particularly in the subset of patients with diabetes, long lesions or small vessel disease.Drug-eluting stents (DES) were developed as a viable method for focused delivery of anti-restenosis compounds to target lesions for the reduction of restenosis. Of the DES available and with the results of up to six (6) years clinical follow-up, the sirolimus-eluting stent (SES) has become the current gold standard for stent implantation. With the advent of using DES to treat complex lesions such as longer lesions requiring the use of multiple stents and the use in bifurcation lesions, the risk of stent thrombosis has increase.Late stent thrombosis has also been reported following DES implantation.Long term treatment with dual anti-platelet therapy following stent implantation has become the solution used to counteract the risk of stent thrombosis, this solution does not come without it's own risks and is an expensive therapy. Another specific problem of DES is delayed endothelization, and this may be and attributing factor in prolonging the period of thrombotic risk as shown by pathological findings at autopsy following SES implantation. These examinations have shown that even after 16 months, neointimal healing is still incomplete with approximately 20% of stent struts being found uncovered. Questions have arose that the problems of late thrombosis and delayed endothelization of stent struts with DES could be the result of the permanent polymer that is used as the bonding agent for the anti-restenosis compounds to the stents.Intravascular Ultrasound (IVUS) along with angiography has been the techniques used to gain data on DES to this point. Angiography is a 2 dimensional tool that gives a view of the vessel and IVUS gives a more 3 dimensional view of the vessel. IVUS does have its limitations, as stent struts are reflectors of sonic waves, shadowing around and behind the struts occurs. IVUS is also limited in detecting malapposition of the struts to the vessel wall especially if the area between the vessel wall and the strut in very small.

RATIONALE Optical Coherence Tomography (OCT) is an optical analogue of IVUS that uses an infrared light source and measures the backscatter of the light. With this technique a higher level of resolution compared with IVUS has been reported.OCT has been reported as being able to visualize and detect atherosclerotic plaques and assess more accurately strut malapposition and the presence or thickness of neointimal hyperplasia as compared to IVUS. With the question of delayed endothelization due to the permanent polymer being a probable risk for late stent thrombosis, it is felt that OCT post stent implantation may give a more accurate assessment of stent strut endothelial coverage.

This study is designed to compare the intimal hyperplasia following implantation of the Excel DES with a biodegradable polymer vs. the Cypher DES with a permanent polymer using OCT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 75 years.
* Binary stenosis of > 70% in a de novo lesion in native coronary artery.
* Reference lumen diameter proximal to the target lesion is 2.5 mm and < 4.0 mm.
* Reference lesion length of < 30 mm.
* The target lesioin can be covered with a makimum of two overlapping stents at a single lesion.
* Written informed consent has been signed.

Exclusion Criteria:

* Pregnant or breast feeding woman.
* Intolerance to aspirin, clopidogrel (Plavix®), ticlopidine(Ticlid®), heparin, bivalirudin, stainless steel, contrast agent(that cannot be adequately premedicated), parylene, poly-lacticacid (PLA), or Biolimus A9 (or its analogues).
* Lesion located in a protected or unprotected Left Main Coronary Artery.
* STEMI within 72 hours prior to index procedure.
* The patient has had another drug-eluting stent (DES) implanted within 12 months prior to the index procedure.
* CCS Class III patients or the patient has a LVEF of < 40%.
* Diffuse lesions of > 40 mm in length.
* Renal impairment, with a serum creatinine of > 2.0 mg/dl.
* Complicated anatomy such as Chronic Total Occlusion (CTO),Bifurcation Lesions (with side branch of > 2.5 mm) or Triple Vessel Disease (TVD).
* Lesion cannot be pre-dilated successfully.
* History of gastritis and/or bleeding history which will limit the usual dual anti-platelet regime.
* Patient has a co-morbid condition(s) that could limit his/her ability to participate in the study, comply with follow-up requirements and impact the scientific integrity of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intends to enroll up to 100 patients from a single center in China. Patients will be randomized in a 1:1 fashion, Excel DES:Cypher DES.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To quantitate the presence of neointimal stent strut coverage at 6 month via Optical Coherence Tomography follow-up. | 6 month

SECONDARY OUTCOMES:
1.Stent strut apposition at 6 month follow-up. 2. Neointimal thickness at 6 month follow-up. 3. late loss at 6 months 4. Major Adverse Cardiac Events | 12 month